CLINICAL TRIAL: NCT02835963
Title: Predictive Criteria of Acute Heart Failure (AHF) in Patients Admitted to Emergency Department for Dyspnea.
Brief Title: Acute Heart Failure Study in Patients Admitted to Emergency Department for Dyspnea
Acronym: PREDICA
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC/31/15/7672
Record Dates: First submitted 2016-07-07; First posted 2016-07-18 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
Keywords: acute heart failure; dyspnea; predictive value
MeSH Terms: conditions — Heart Failure; Dyspnea | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Data collection — Usual data collection

SUMMARY:
No studies have analyzed the predictive value of different anamnestic and clinical signs for the diagnosis of acute heart failure (AHF) in patients admitted to emergency department. That's why the expert group of the AHF of South West of France mobilizes to conduct this study to evaluate the diagnostic predictive value of different anamnestic and clinical signs for the diagnosis of AHF to emergencies.

DETAILED DESCRIPTION:
There is no recommendation of the French Society of Emergency Medicine (SFMU) on the management of the acute heart failure in the emergency department.

The present study hypothesizes that identifying anamnestic and clinical criteria of AHF in patients admitted to emergency department for acute dyspnea would optimize the management of these patients upon arrival to the emergency department and to implement rapidly the appropriate therapeutic strategies.

All patients admitted for dyspnea will be enrolled by the emergency physicians (after verification of inclusion and exclusion criteria) in the 3 participating centers.

Then, all files will be analyzed retrospectively from information collected by a committee of experts cardiologists and emergency physicians of each center.

The primary objective is the evaluation of diagnostic predictive value of different anamnestic and clinical signs for the diagnosis of AHF in emergency department for the construction of a clinical prediction score of acute heart failure. The secondary objective is the description of the diagnostic and therapeutic management of patients admitted to the emergency for acute dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years
* Admitted to emergency department for acute dyspnea

Exclusion Criteria:

* Traumatic dyspnea
* shock / Systolic blood pressure <90 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from which the cohort will be selected is patients admitted to hospital center emergency department of Toulouse, Bordeaux and Pau.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
diagnosis of AHF after expertise | 12 months
  The final diagnosis of AHF after expertise of patients records by a committee of experts cardiologists and emergency physicians.

SECONDARY OUTCOMES:
Diagnostic and therapeutic management of patients admitted to the emergency for acute dyspnea | Baseline
  The secondary objective is the description of the diagnostic and therapeutic management of patients admitted to the emergency for acute dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: CHARPENTIER Sandrine, MD PhD, Principal Investigator — University Hospital, Toulouse; RONCALLI Jérome, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - University Hospital, Bordeaux
  - Hospital, Pau
  - University Hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Roncalli J, Picard F, Delarche N, Faure I, Pradeau C, Thicoipe M, Galinier M, Charpentier S. Predictive criteria for acute heart failure in emergency department patients with acute dyspnoea: the PREDICA study. Eur J Emerg Med. 2019 Dec;26(6):400-404. doi: 10.1097/MEJ.0000000000000622. PMID 31453847